CLINICAL TRIAL: NCT07271017
Title: Robot-Assisted Prostate Biopsy With a Novel Ultrasound Probe
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB00229568; R01CA303859 (NIH)
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer (Diagnosis)
Keywords: Robot biopsy; Fusion biopsy; MRI targeted biopsy; Systematic biopsy; Personalized biopsy; Precision biopsy; Biopsy optimization
MeSH Terms: conditions — Prostatic Neoplasms; Disease

STUDY DESIGN:
Intervention Model Description: Patients are enrolled consecutively in the TR or TP biopsy groups by the urologists and accounting for patient's preference
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Transrectal biopsy (TR) (Experimental): Biopsy guided by transrectal ultrasound fused with MRI and needle inserted on a transrectal path
  Interventions: Device: Prostate biopsy
- Transperineal biopsy (TP) (Experimental): Biopsy guided by transrectal ultrasound fused with MRI and needle inserted on a transperineal path.
  Interventions: Device: Prostate biopsy

INTERVENTIONS:
Device: Prostate biopsy — Precision personalized prostate biopsy with a novel ultrasound probe and robot, ProBot

SUMMARY:
Prostate cancer (PCa) is the most diagnosed type of cancer and the second leading cause of cancer related deaths among US men, and its incidence has increased steadily in the last decade. Efforts to address the rise in PCa diagnosis without overdetection and overtreatment include targeted biopsy techniques for clinically significant PCa using magnetic resonance imaging (MRI), and precision targeted biopsy guided by ultrasound and fused to the MRI.

The study aims to improve prostate biopsy with a novel ultrasound probe and robot developed at Johns Hopkins, the ProBot device. The trial is a Phase 1 clinical trial to evaluate the safety and feasibility of the new device.

ProBot is an entirely new concept including a novel ultrasound probe and robot kinematics specifically designed for the prostate. It operates with only two degrees of freedom configured such that the motions for 3D image scanning and biopsy may not deform the prostate gland, thus improving the accuracy of MRI-ultrasound fusion and needle targeting at biopsy.

ProBot is a small and lightweight robot (1.3Kg including the ultrasound probe). It allows hands-free operation of its ultrasound probe at 3D image scanning and needle targeting supervised by the urologist.

In addition to MRI-targeted biopsy (TB), at systematic biopsy (SB), instead of using the common template plan that is the same for all patients, the innovative software optimizes the plan for each patient to obtain a diagnosis that is representative of the whole gland histology. The ProBot robot is also uniquely capable of transrectal (TR) and transperineal (TP) biopsy.

The aims of the study are to determine the safety and feasibility of the new device at TR and TP biopsies.

ELIGIBILITY:
Included in the study will be:

* Men between the ages of 40 and 75
* Men must have one of the following "high risk" features:

  1. PSA > 4.0 ng/ml and/or abnormal digital rectal examination (DRE)
  2. ASAP (atypical small acinar proliferation) on previous biopsy
* Men with mpMRI or bpMRI exams, including both PI-RADS ≤2 and PI-RADS ≥3.

Excluded from the study will be patients without available mpMRI exams and patients:

* Females and children because of the prostate cancer targeted disease.
* Patients who are not recommended or in whom TR or TP prostate biopsy is considered high-risk:

  1. Patients with previous rectal surgery.
  2. Patients with anal stenosis or coagulopathy.
  3. Patients on active anticoagulation medication (eg. Coumadin, Lovenox, or Heparin).
  4. Patients who cannot tolerate periprostatic Lidocaine block anesthesia or in whom anesthesia is considered high-risk.
* Patients who already had a prostate biopsy taken with the ProBot investigational device.
* Vulnerable populations, such as prisoners, institutionalized individuals.
* Patients who are unwilling or unable to sign informed consent (no assent required).

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2030-05-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Device feasibility as assessed by patient discomfort score | Immediately after the procedure
  Scale 1-10, 10 highest discomfort
Device feasibility as assessed by maximal procedural pain | Immediately after the procedure
  Scale 1-10, 10 highest pain
Device feasibility as assessed by the rate of complications | Throughout the study, each case recorded within 1 month of the procedure
  Rate of complications
Device feasibility as assessed by serious adverse events | Up to 1 month post procedure
  Serious Adverse events throughout the study
Device feasibility as assessed by the rate of successful completion of cases | Immediately post procedure
  Rate of cases completed successfully throughout the study
Device feasibility as assessed by the procedure time | Immediately post procedure
  Times of the procedures measured in minutes throughout the study

SECONDARY OUTCOMES:
Prostate cancer detection rates at targeted biopsy (TB) | Up to 1 month post procedure
  Clinically significant PCa detection rates at TB throughout the study
Prostate cancer detection rates at systematic biopsy (SB) | Up to one month post procedure
  Clinically significant PCa detection rates at SB throughout the study
Needle targeting errors | Immediately post procedure
  Measured in ultrasound throughout the study
Prostate deformations (mm) | Immediately post procedure
  Maximum deformation of the gland between the start and end of the procedure measured in [mm] throughout the study
Prostate displacement (mm) | Immediately post procedure
  Displacement of the gland between the start and end of the procedure measured in [mm] throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Misop Han, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No